CLINICAL TRIAL: NCT06610435
Title: Effects of Manual Therapy and Home Exercise Treatment on Pain, Stress, Sleep and Life Quality in Patients with Bruxism: a Randomized Clinical Trial
Brief Title: Effects of Manual Therapy and Home Exercise in Bruxism
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ankara University (Other)
Responsible Party: Principal Investigator, Merve Berika Kadıoğlu, Lecturer, Ankara University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2024-SBB-0289
Record Dates: First submitted 2024-09-18; First posted 2024-09-24 (Actual); Last update posted 2024-09-24 (Actual); Status verified 2024-09

CONDITIONS: Bruxism; Manual Theapy; Exercise; Orofacial Pain
Keywords: Manual Therapy; Exercise; Physiotherapy; Bruxism; Sleep and Life Quality
MeSH Terms: conditions — Bruxism; Motor Activity; Facial Pain | interventions — Musculoskeletal Manipulations

STUDY DESIGN:
Intervention Model Description: Thirty patients with bruxism were randomly divided into as Manual Therapy Group (15) and Home Exercise Group (15).
Who Masked: Outcomes Assessor
Masking Description: To ensure blinding, baseline and final outcome measurements were performed by researchers other than the physiotherapist performing manual therapy.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Manual Therapy (Experimental): The term manual therapy includes a wide variety of detailed applications ranging from joint-oriented applications (joint mobilizations and/or manipulations) or soft tissue techniques (muscle stretching or trigger point therapy) to therapeutic exercises. Manual therapy in our study was used to restore normal temporomandibular joint range of motion, reduce local ischemia, stimulate proprioception, break fibrous adhesions, stimulate synovial fluid production and reduce pain.
  Interventions: Procedure: Manual Therapy
- Home Exercise (Experimental): Exercise therapy, one of the physical therapy applications, has an important place in the rehabilitation of musculoskeletal disorders. With this method, it is aimed to decrease inflammation, increase coordination of muscle activity, promote tissue repair and regeneration, relieve pain and restore normal function. In addition to the special exercises known as Rocabado exercises which are used in the treatment of temporomandibular joint, various studies have been performed in which mobilization, coordination, posture and relaxation exercises were used for the treatment of disorders related to the masticatory system and it has been emphasized that studies on this subject should be continued.
  Interventions: Procedure: Home Exercise

INTERVENTIONS:
Procedure: Manual Therapy — Various soft tissue and joint mobilizations, intramuscular stretches, trigger point treatments, and intraoral applications for the temporomandibular joint were performed in 15 randomly selected bruxism patients. Soft tissue mobilization techniques were applied bilaterally on the trigger points in the masseter, temporal, lateral and medial pterygoid muscles of the masticatory muscles in the transverse direction from inside and outside the mouth. In addition, deep friction massage and myofascial relaxation techniques were applied to suprahyoid and infrahyoid muscles, sternocleidomastoid, scalene, upper trapezius, levator scapula and suboccipital muscles until relaxation was felt. In addition, distraction and bridging techniques were applied in the suboccipital region to release the tissue and fascia techniques were applied in the cervical region to loosen the fascia. The manual therapy procedure, which was applied in the supine position and lasted approximately 40 minutes for 8 weeks
  Arms: Manual Therapy
Procedure: Home Exercise — The exercise group consisted of 15 randomly selected bruxist individuals and aimed to reduce pain, decrease involuntary contractions of masticatory muscles, increase their nutrition, flexibility and coordination, and strengthen weak muscles with exercise therapy. These exercises consist of resistant isometric jaw movements to increase coordination and relaxation of the masticatory muscles (post isometric relaxation technique), Rocabado exercises, stretching and posture exercises for temporal, masseter and suprahyoid muscles as well as neck muscles. All individuals in this group were taught the programmed exercises practically and were asked to repeat the home exercises (lasting approximately 25 minutes) three times a week for 8 weeks. In addition, a video explaining the exercises in detail was shared with all participants in the group in order to ensure that the exercises were not forgotten and to achieve accuracy and standardization among the participants.
  Arms: Home Exercise

SUMMARY:
Objectives: This trial aimed to examine the effects of manual therapy and home exercise treatments on pain, sleep quality, stress level and quality of life in patients with bruxism.

Methods: Thirty bruxists over the age of 18 were included in the study. The patients were randomly divided into Manual Therapy Group (MTG) and Home Exercise Group (HEG). Before treatment (T1) demographic information was obtained from all patients, they were asked to fill out the Pittsburgh Sleep Quality Index (PSQI), Perceived Stress Scale (PSS), Fonseca Anamnestic Index (FAI) and Quality of Life Scale/Short Form-36 (SF-36) and number of trigger points and pain levels were determined at baseline. Manual therapy and home exercises were applied to both groups for 8 weeks and all tests were repeated and re-evaluated at the end of 8 weeks (T2). After that, the data was analyzed with statistical tests.

DETAILED DESCRIPTION:
Bruxism is a common parafunctional habit defined as clenching and/or grinding of teeth occurring during sleep and/or wakefulness. Although the etiology is not known exactly, there is a consensus that it is multifactorial. Emotional stress is one of the important factors leading to bruxism. It has been shown that a stressful life has an important effect in explaining clenching during the day. In addition to stress, previous studies showing that psychiatric disorders, especially depression and anxiety disorders, accompany TMD and bruxism.

This trial aimed to examine the effects of manual therapy and home exercise treatments on pain, sleep quality, stress level and quality of life in patients with bruxism. In the study thirty bruxists over the age of 18 were included in the research protocol. The patients were randomly divided into Manual Therapy Group (MTG) and Home Exercise Group (HEG). Before treatment (T1) demographic information was obtained from all patients, they were asked to fill out the Pittsburgh Sleep Quality Index (PSQI), Perceived Stress Scale (PSS), Fonseca Anamnestic Index (FAI) and Quality of Life Scale/Short Form-36 (SF-36) and number of trigger points and pain levels were determined at baseline. Manual therapy and home exercises were applied to both groups for 8 weeks and all tests were repeated and re-evaluated at the end of 8 weeks (T2). The normal distribution of the groups was tested with Kolmogorov-Smirnov. Paired Samples t test was used for intra-group comparisons at T1 and T2, and Independent t test was used for inter-group comparisons. The statistical significance level was accepted as p<0.05.

ELIGIBILITY:
Inclusion Criteria:

* Volunteer students aged between 18-25
* Answered "yes" to at least two of the six questions in the Bruxism questionnaire.

Is there anyone hear you grinding your teeth at night? Do you feel fatigue or pain in your jaw when you wake up in the morning? Do you feel pain in your teeth and gums when you wake up in the morning? Do you have a headache when you wake up in the morning? Do you notice that you grind your teeth during the day? Do you notice that you clench your teeth during the day?

- Having at least two clinical signs of bruxism Abnormal tooth wear on the occlusal surfaces of the teeth Abfraction Gingival recession and/or cervical defect Tongue indentations or damage to the inside of the cheek Tense facial and jaw muscles, muscle sensitivity, and masseteric hypertrophy upon bidigital palpation

Exclusion Criteria:

* Characterized by a neurological disease,
* Botulinum toxin injections into the masticatory muscles in the last year,
* Using antidepressant-type medications that will affect the central nervous system,
* Receiving occlusal splint treatment,
* Having more than two molar teeth missing in the posterior

Ages: 18 Years to 25 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 30 (Actual)
Dates: Start 2024-05-01 (Actual); Primary Completion 2024-08-20 (Actual); Study Completion 2024-08-25 (Actual)

PRIMARY OUTCOMES:
Pain Level | From baseline to the end of treatment at 8 weeks
  Visual analog scale (VAS) was used to assess the severity of pain related to bruxism. On a 10 cm long horizontal line, "0 (no pain)" was written at the beginning and "10 (most intense pain)" was written at the end and the patient was asked to mark the pain intensity they perceived at rest, active use and at night on the line. The pain intensity of the individual was recorded by measuring the distance marked on the line in millimeters. It has been reported that the Turkish version of the VAS is a valid and reliable measurement tool in the evaluation of musculoskeletal disorders
Sleep Quality Index | From baseline to the end of the treatment at 8 weeks
  It was examined with Pittsburgh Sleep Quality Index (PSQI). It is a 24-question scale developed by Buysse et al. in 1989 that evaluates sleep quality in the last month, and the last 5 questions are used only for clinical evaluation. The sum of the scores of 7 components including subjective sleep quality, sleep latency, sleep duration, habitual sleep efficiency, sleep disturbance, sleep medication use and daytime dysfunction gives the total score index. The total PDQI score ranges from 0 to 21; a score above 5 points indicates poor sleep quality; a score of 5 points or less indicates good sleep quality.
Stress level | From baseline to the end of the treatment at 8 weeks
  It was examined with Perceived Stress Scale.It was developed by Cohen, Kamarck and Mermelstein (1983) and consists of 14 items. The scale consists of two sub-dimensions: stress/discomfort perception and self-efficacy perception. Participants rate the stress they perceive in the scale as "0" never, "1" almost never, "2" sometimes, "3" often, and "4" very often. The stress level perceived by individuals is determined by summing the scores obtained from the items. A score between 0-56 points is obtained from the scale and the higher the score, the higher the perceived stress level.
Quality of Life | From baseline to the end of the treatment at 8 weeks
  It was examined with Short Form-36 (SF-36) Quality of Life Scale. SF-36 was developed by the Rand Corporation to obtain information about the health status of the individual. It consists of 8 sub-dimensions and 36 items. The sub-dimensions consist of physical function, social function, physical role difficulty, emotional state difficulty, mental health, energy/vitality, pain, and general perception of health. "0" represents the worst health status, while "100" represents the best health status. Each sub-dimension is evaluated individually without calculating the total score, and in our study, general health perception was evaluated.

SECONDARY OUTCOMES:
Presence and severity of Temporomandibular Joint Disorder (TMD) symptoms | From baseline to the end of the treatment at 8 weeks
  It was examined with Fonseca Anamnestic Index (FAI). It was developed in 1994 by Fonseca et al. and consists of 10 questions investigating pain in the head and TMJ (Table 2.) The questionnaire includes various questions about joint, head and neck pain, joint movements, parafunctional habits, impaired occlusion and emotional stress. Participants were asked to answer 'Yes' (10 points), 'No' (0 points) and 'Sometimes' (5 points) to each question and TMD was classified as none, mild, moderate and severe according to the total score.
Bruxism | From baseline to the end of the treatment at 8 weeks
  It was examined with Bruxism Questionnaire. According to the survey questions prepared by referencing the studies of Pintado et al and Shetty et al, it was stated that individuals who answered "Yes" to at least two of the questions specified in the survey can be called bruxists. The total score range varies between 0-6.
Trigger Point | From baseline to the end of the treatment at 8 weeks
  While evaluating the trigger points in the masticatory and neck muscles, the tense muscle was palpated with a fingertip. Palpation was performed along the long axis of the tense muscle and the most sensitive point was determined. Sudden reaction or vocal response of the patient with light pressure applied to this point and the presence of reflected pain in a region distant from this region indicated the presence of a trigger point. Evaluation was performed in 14 muscles and the muscles with trigger points and the total number of trigger points were recorded.

CONTACTS AND LOCATIONS:
Locations (1):
- Ankara University, Faculty of Dentistry, Ankara, Emniyet, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Yes
We can share the questionnaires and indexes used in the study
Supporting Information: Study Protocol